CLINICAL TRIAL: NCT02034045
Title: The Expanding Paramedicine in the Community (Study)
Brief Title: Expanding Paramedicine in the Community
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EPIC - RCT
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus (DM); Congestive Heart Failure (CHF); Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Active Comparator): Patients randomized to the control group will continue to receive usual care from their Family Health Care Team. Usual care includes physician assessment and treatment and periodic augmentation of care in the community (CCAC or case manager, nurse practitioner) at the discretion of the treating physician.
  Interventions: Other: Usual Care
- Community Paramedicine (Experimental): The intervention will consist of an initial visit and 3 follow-up visits at 3 month intervals over one year by a paramedic who has received additional training in chronic disease management, in addition to routine usual care and any additional visits prompted by the patient, the paramedic or the Family Health Care Team.
  Interventions: Other: Community Paramedicine

INTERVENTIONS:
Other: Community Paramedicine
  Arms: Community Paramedicine
Other: Usual Care
  Arms: Usual Care

SUMMARY:
Initiatives aimed at reducing Emergency Department (ED) wait times and improved community health initiatives are major priorities in Canada. Three of the most common chronic diseases worldwide are Diabetes Mellitus (DM), Congestive Heart Failure (CHF) and Chronic Obstructive Pulmonary Disease (COPD). These diseases are on the rise and currently cost the Canadian health care system billions of dollars every year including the cost of hospitalizations and ED visits. The existing health care system does not have the resources and manpower to effectively care for these patients in the future.

Paramedics are currently employed to provide Emergency Medical Services in remote, rural and urban settings in Canada.

They are highly trained health care practitioners that are mobile in the community and currently work in a physician medically delegated act model and therefore are positioned to take on new collaborative roles to deliver patient care in the community setting. Increased community paramedic care could decrease the utilization of the health care system resources for patients with chronic disease. Using a randomized control trial design we will attempt to answer the question of whether whether non-emergency community paramedics conducting home visits to undertake assessments and evidence-based treatments of patients in partnership with family doctors will decrease the rate of patient hospitalization.

DETAILED DESCRIPTION:
Imagine if we could leverage existing infrastructure to enhance how we better manage and support patients with chronic disease in the community? Three of the most common chronic diseases worldwide are Diabetes Mellitus (DM), Congestive Heart Failure (CHF) and Chronic Obstructive Pulmonary Disease (COPD). These diseases are on the rise and currently cost the Canadian health care system billions of dollars every year including the cost of unnecessary hospitalizations and ED visits. The current structure of the health care system does not have the capacity to effectively care for these patients in the future. Paramedics are currently employed 24-7 to provide Emergency Medical Services (EMS) in urban, rural and settings across Canada. They are highly trained health care practitioners that are connected to and mobile in the community and currently work in a medically delegated act model with physicians where they regularly rely on independent judgment giving them a significant advantage in assessing patients. The evidence already tells us that collaborative Chronic Care Models can improve patient outcomes and decrease overall health care utilization. What if we leveraged this incredible resource to enhance patient care in the community setting? We hypothesize that training paramedics in chronic disease management and having them conduct home visits to assess and treat patients under medical delegation of the patients' primary care physicians will reduce the rate of acute care hospitalization and, ED visits, EMS utilization, and Family Health Team (FHT) utilization for COPD, DM and CHF patients.

So how do we find out if it works? We propose a randomized controlled trial (Level 1 evidence) to rigorously study the effectiveness of community paramedicine model versus standard care. The primary study question is whether non-emergency community paramedics conducting home visits to undertake assessments and evidence-based treatments of patients under the medical delegation of primary care physicians will decrease the rate of hospitalization for chronic disease patients. Our intervention will be applied in select Ontario Family Health Team (FHT) patients diagnosed with COPD, CHF and DM. We plan to randomize 695 patients: patients randomized to the intervention group will be assessed and treated during home visits by community paramedics. Patients randomized to the control group will continue to receive usual care from the participating Family Health Teams. The number of hospitalizations, hospital length of stay, ED visits, EMS utilization and cost-effectiveness will be compared using existing administrative databases. We have been doing a feasibility trial since March of 2013 to confirm our recruitment and data collection approaches.

The intent of the Partnerships for Health System Improvement (PHSI) program is to strengthen Canada's health care system through collaborative, applied and policy-relevant research. Our project has been developed in strong partnership with Centennial College; Central Community Care Access Centre; York Region Emergency Medical Services; Health For All Family Health Team; Markham Family Health Team; Rescu, Li Ka Shing Knowledge Institute, St. Michael's Hospital; and the Sunnybrook Centre for Prehospital Medicine. We have also partnered directly with the Primary Care Branch of the Ministry of Health and Long Term Care to ensure a fruitful integrated knowledge translation plan at the policy level. By engaging all of the key stakeholders upfront we have already created the necessary linkages to make this health system innovation possible.

If found to be effective, the simplicity of the community paramedicine model allows it to be scalable in various ways for EMS services across the country. It could also be expanded to include management of several other conditions. Funding is only getting tighter and health care capacities will be increasingly challenged in the coming years - innovation in how we use existing resources is the future of health system improvement. Community paramedicine is a perfect example of this type of innovation and our project will provide the evidence needed by decision makers and knowledge users to significantly impact primary care policy making for the future.

ELIGIBILITY:
Inclusion Criteria:

Residents of the region of York, Ontario, 18 years of age or older, diagnosed at any point in time with COPD, CHF, or DM and identified by the Family Health Care Team as high risk for admission.

Exclusion Criteria:

Residents of long-term care facilities or if have cognitive impairment, uncontrolled psychiatric disease or language barriers that would make it difficult to understand the consent and communicate with the paramedic during the scheduled visits, unless the individual with power of attorney for personal care consented and agreed to be at each visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Hospital admissions per patient | maximum 2 years
  The primary outcome of this trial is the one-year measurement of hospital admissions per patient.

SECONDARY OUTCOMES:
Health Resource Utilization | maximum 2 years
  The secondary outcomes will be measures of health system utilization at one year (reported as all cause and disease specific) and will include:
  1. Calls to 911 (regardless of whether patient was transported to hospital)
  2. Visits to the participating Family Health Team clinics and any after-hours clinics
  3. Length of stay in hospital
Cost Effectiveness | maximum 2 years
  Cost effectiveness analysis for this model of care based on the composite outcome measures.

OTHER OUTCOMES:
Trial Fidelity and Safety | maximum 2 years
  Measures of intervention compliance and safety (ie. Completed assessments and visits, protocol violations identified by physician review of EMR)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Morrison, MD, MSc, FRCPC, Principal Investigator — Unity Health Toronto
Locations (4):
- Canada (4):
  - Health for All and Markham Family Health Team, Markham, Ontario
  - Aurora-Newmarket Family Health Team, Newmarket, Ontario
  - Owen Sound Family Health Team, Owen Sound, Ontario
  - Stouffville Medical Centre, Stouffville, Ontario

REFERENCES:
- [Derived] Poot CC, Meijer E, Kruis AL, Smidt N, Chavannes NH, Honkoop PJ. Integrated disease management interventions for patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2021 Sep 8;9(9):CD009437. doi: 10.1002/14651858.CD009437.pub3. PMID 34495549
- [Derived] Heinelt M, Drennan IR, Kim J, Lucas S, Grant K, Spearen C, Tavares W, Al-Imari L, Philpott J, Hoogeveen P, Morrison LJ. Prehospital Identification of Underlying Coronary Artery Disease by Community Paramedics. Prehosp Emerg Care. 2015;19(4):548-53. doi: 10.3109/10903127.2015.1005261. Epub 2015 Apr 24. PMID 25909892
- [Derived] Drennan IR, Dainty KN, Hoogeveen P, Atzema CL, Barrette N, Hawker G, Hoch JS, Isaranuwatchai W, Philpott J, Spearen C, Tavares W, Turner L, Farrell M, Filosa T, Kane J, Kiss A, Morrison LJ. Expanding Paramedicine in the Community (EPIC): study protocol for a randomized controlled trial. Trials. 2014 Dec 2;15:473. doi: 10.1186/1745-6215-15-473. PMID 25467772